CLINICAL TRIAL: NCT00837239
Title: A Randomized, Placebo-controlled, Blinded Phase II Study of Huachansu & Gemcitabine in Pancreatic Cancer
Brief Title: Huachansu & Gemcitabine in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-0948
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Pancreatic Cancer
Keywords: HuaChanSu; HCS; Gastrointestinal; Gastrointestinal Disease; Metastases; Cancer; Pancreatic cancer; Placebo; Gemcitabine; Gemcitabine Hydrocholoride; Gemzar; Fudan UniversityCancer Hospital
MeSH Terms: conditions — Pancreatic Neoplasms; Gastrointestinal Diseases; Neoplasm Metastasis; Neoplasms | interventions — Gemcitabine; huachansu

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine + HuaChanSu (Experimental): Gemcitabine 1,000 mg/m2 once a week for 3 weeks then 1 week off + HuaChanSu 20 mL/m2 for total 500 mL given as a 2 hour infusion, 5 days a week for 3 weeks then one week off (28 Day Cycle).
  Interventions: Drug: Gemcitabine; Drug: HuaChanSu
- Gemcitabine + Placebo (Experimental): Gemcitabine 1,000 mg/m2 once a week for 3 weeks then 1 week off (28 Day Cycle) + Placebo 500 ml saline only administered as a 2 hour infusion by central line.
  Interventions: Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Gemcitabine — 1,000 mg/m2 once a week for 3 weeks then 1 week off (28 Day Cycle).
  Other Names: Gemcitabine Hydrocholoride; Gemzar
Drug: HuaChanSu — 20 mL/m2 for total 500 mL given as a 2 hour infusion, 5 days a week for 3 weeks then one week off (28 Day Cycle).
  Other Names: HCS
  Arms: Gemcitabine + HuaChanSu
Drug: Placebo — 500 ml saline only administered as a 2 hour infusion by central line.
  Arms: Gemcitabine + Placebo

SUMMARY:
This protocol is part of a larger grant funded by the NCI to create an international research center to study traditional Chinese medicine (TCM). All of the patients enrolled in this study will be treated at the Cancer Hospital, Fudan University, our sister institution in Shanghai, China. No patients will be seen at MDACC. This protocol will be overseen by the Fudan University Institutional Review Board (IRB00002408) which has Federal Wide Assurance through the U.S. Department of Health & Human Services (Approved: April 25, 2002). The research nurses have received training at MDACC and will receive regular oversight by MDACC personnel.

Primary End Point:

1. Determine the efficacy of huachansu as measured by progression free survival at 4 months.

Secondary End Points:

1. Examine the feasibility and safety of treatment using huachansu in combination with gemcitabine in patients with pancreatic cancer.
2. Determine clinical efficacy by other measures including tumor response, 6-month survival, and changes in quality of life (QOL) in patients with pancreatic cancer.
3. Monitor patient blood levels of the three main cardiac glycosides that are in huachansu (bufalin, cinobufagin, and resibufogenin). This information will provide evidence to delineate the role of these cardiac glycosides in antitumor activity.

DETAILED DESCRIPTION:
The Study Drugs:

HuaChanSu is a substance used in China to treat different types of cancer. One of the major elements of the substance is bufalin, which is an ingredient that has been shown to block the growth of tumor cells.

Gemcitabine is designed to disrupt the growth of cancer cells, which may cause cancer cells to die.

Screening:

Before you can receive study treatment, you will have "screening tests." These tests will help the study doctor decide if you are eligible to take part in this study. The following tests will be performed:

* You will be asked questions about your medical history and any symptoms you may have now.
* You will have a complete physical exam.
* Your vital signs (temperature, heart rate, breathing rate, and blood pressure), height, and weight will be measured.
* You will be asked how well you are able to perform the normal activities of daily living (a performance status evaluation).
* You will have an electrocardiogram (ECG-a test that measures the electrical activity of the heart).
* To check the status of the cancer, you will have computed tomography (CT) scan(s) and/or magnetic resonance imaging (MRI) scans of your abdomen, pelvis, and any other areas where there is disease.
* You will complete a short questionnaire that will ask questions about your quality of life. This will take about 5 minutes to complete.
* A traditional Chinese medicine diagnosis will also be done. This will include diagnosis by a study doctor. The doctor will take your pulse (heart rate), look at your tongue, and ask you a few questions about your health. The doctor will also use a heart-rate machine and take a photograph of your tongue. This will allow a more scientific check of your heart rate and tongue condition.
* You will have blood (about 3 teaspoons) collected for routine safety tests. This routine blood draw will include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative.
* You will have 1 biopsy of your tumor tissue to check your cancer type. To collect a tumor tissue biopsy, an area where cancer is located is numbed with anesthetic, and a small amount of tumor tissue is withdrawn through a large needle.

Randomization:

If you are found to be eligible and decide to take part in this study, you may begin treatment.

The first 3 participants enrolled on this study will be given HuaChanSu and gemcitabine, to find out if this dose combination can be tolerated. After the first 3 participants are enrolled, all other participants will be randomly assigned (as in the toss of a coin) to receive HuaChanSu and gemcitabine or gemcitabine and the placebo. The first 20 participants have an equal chance of receiving HuaChanSu or placebo, but after that point, participants will have a better chance of being assigned to the group that is responding better to their study combination. All participants will receive the same dose level of gemcitabine, but you will not know if you are given HuaChanSu or placebo. However, this information can be found out if medically necessary.

Study Treatment:

Before the study drug infusions begin, you will be fitted with a peripherally-inserted central catheter (PICC) by a specially trained nurse. A PICC is a tube that is inserted into a vein, either in your arm or under the collarbone, to make it easier to give you gemcitabine with or without HuaChanSu. This is an outpatient procedure. You will be given a separate consent form for the insertion of the PICC. It will explain the risks of the procedure and how to take care of the PICC. Your doses of gemcitabine and either HuaChanSu or a placebo (a saline [salt water] solution that looks like HuaChanSu but has no effects) will be given through the PICC while you are on this study.

* HuaChanSu (or placebo) will be given as a 2-hour continuous (nonstop) infusion through the PICC. You will receive the 2-hour dose 5 days a week (5 days in a row each time) for 3 weeks. This will be followed by 1 week of not receiving the drug.
* Gemcitabine will be given through a needle in a vein over 30 minutes on Days 1, 8, and 15, followed by 1 week where no study drug is given. Each 4-week treatment period is called a study "cycle."

PK Testing:

During Cycle 1 only, you will have extra blood (about 1 teaspoon each time) collected at various time points for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points. PK blood samples will be drawn 4 times over a 24-hour period on Day 1 and then once each on Days 7, 14, and 21.

Study Tests:

Before each new cycle, you will be asked questions about your current health, and you will have a complete physical exam. Your vital signs and weight will be measured. You will have a performance status evaluation. You will complete a questionnaire about your quality of life. The questionnaire will take about 5 minutes to complete. You will also have blood (about 3 teaspoons) drawn for routine safety tests.

On Days 8 and 15 of each cycle, you will also have blood (about 3 teaspoons) drawn for routine safety tests.

Every 8 weeks (starting in Cycle 3), to check the status of the cancer, you will have CT and/or MRI scan(s) of your abdomen, pelvis, and any other areas where there is disease.

Length of Study Participation:

You may continue to receive more cycles of treatment, as long as the cancer does not get worse and intolerable side effects do not occur.

You will be taken off this study if the cancer gets worse, intolerable side effects occur, new information shows that the treatment is not right for you, you are not able to follow the study rules, the study is stopped, or you decide to leave the study for any reason. If you are thinking about leaving the study, please tell your study doctor, so that you may be told how to end treatment safely as well as what other treatment options are available.

End-of-Treatment Visit:

You will be asked to have a final study visit 4 weeks after your last dose of study drugs. During this visit, you will have the following tests and procedures performed:

* You will have blood (about 3 teaspoons) drawn for routine safety tests.
* You will be asked questions about your medical history.
* You will have a complete physical exam, and your vital signs and weight will be measured.
* You will have a performance status evaluation.
* You will complete a questionnaire about your quality of life.
* To check the status of the cancer, you will have computed tomography (CT) scan(s) and/or magnetic resonance imaging (MRI) scans of your abdomen, pelvis, and any other areas where there is disease (if these were not performed close to the time that you stopped study treatment).

This is an investigational study. HuaChanSu is a commercially available medication that is approved by the Chinese FDA for the treatment of pancreatic cancer. Gemcitabine is approved by the Chinese FDA for the treatment of pancreatic cancer. In this study, the combination of these drugs is being used for research only.

Up to 80 patients will take part in this study. All will be enrolled at Fudan University Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed unresectable (locally advanced or stage IV) pancreatic adenocarcinoma.
2. Karnofsky Performance Status > 60 (see Appendix H for definition)
3. Measurable disease by RECIST criteria must be present. Bone scan abnormalities alone will not be accepted as measurable disease. Lytic lesions seen on plain radiographs will not be accepted as measurable disease but will be evaluated in conjunction with bone scan abnormalities. Pure blastic bone metastases will not be accepted as measurable disease. Pleural or peritoneal effusions will not be accepted as measurable disease. Irradiated lesions are not considered measurable.
4. Patients must not be pregnant. Serum beta-HCG will be checked in all premenopausal patients.
5. Patients must have adequate organ functions reflected by the laboratory criteria below: Granulocytes >1,500/uL; Hemoglobin >/= 8.0 gm/dL; Platelets > 100,000/uL; Serum creatinine < 2.0 mg/dL; Bilirubin < 1.5 mg/dL; SGPT < 3 x normal; Alk Phos < 3 x normal; Calcium </=11.0 mg/dL
6. Age >/=18
7. Patients must not have received any prior chemotherapy. Prior exposure to Traditional Chinese Medicine is allowed provided that at least one week washout time is given prior to initiation of experimental treatment.
8. Concomitant bisphosphonates are allowed for patients with bone metastases.
9. Patients with jaundice must have a biliary drainage decompression operation before recruitment.
10. Ability to understand and the willingness to sign a written informed consent.
11. Prior local therapy, e.g., TACE or radiation, is allowed provided that at least 4 weeks washout time is given.

Exclusion Criteria:

1. Known central nervous system involvement and leptomeningeal disease
2. Other serious illness or condition including cardiac disease including congestive heart failure (New York Heart Association Classification III or IV), active HIV infection/HIV disease, psychiatric disorders.
3. Known allergies to the huachansu or toad skin products.
4. Concurrent infection requiring intravenous antibiotics.
5. Pregnant or lactating women.
6. Prior treatment with systemic chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival at 4 Months | 4 Months
  Number of participants without disease progression four months following treatment.

SECONDARY OUTCOMES:
Median Overall Survival | Up to 4 Years
  Median participants overall survival defined as date of study entry until death, or censored to last known date of survival, reported in days.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Garrett, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- Cancer Hospital Fudan University, Shanghai, China

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org